CLINICAL TRIAL: NCT01308944
Title: Feasibility Study: Therapeutic Targeting of Stress Factors in Ovarian Cancer Patients
Brief Title: Therapeutic Targeting of Stress Factors in Ovarian Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0447 / 201104047
Record Dates: First submitted 2011-02-16; First posted 2011-03-04 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Invasive Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: invasive epithelial ovarian cancer,; primary peritoneal carcinoma,; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Propranolol 40mg po orally twice daily to begin at least 48 hours prior to surgical debulking. This will ideally be titrated in order to maintain a heart rate between 60 and 80 without hypotension.
  After surgery, the patient will resume the propranolol once tolerating clear liquids in the hospital and will remain on them until completion of chemotherapy.
  After completion of chemotherapy, the patient will be weaned off the medication over the following two weeks.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol
  Other Names: Inderal

SUMMARY:
This research is looking at the effect of biobehavioral factors such as stress and whether these factors alter how the body responds to chemotherapy, one of the purposes of this study is to determine if the addition of a beta-blocker such as Propranolol (Inderal) is tolerable when given with chemotherapy in the treatment of newly diagnosed ovarian, fallopian tube, or primary peritoneal cancer. An additional purpose of the study is to understand if behavioral factors such as depression and anxiety can alter different blood markers that affect tumor vascularity. The Investigator wishes to determine whether the use of beta-blocker drugs such as Inderal, might alter these behavioral factors by drawing blood prior to and after the administration of Inderal as well as giving behavioral questionaires at different time points. Beta-blockers are commonly used for the treatment of hypertension, protection of the heart after a heart attack, and irregularities in heartbeats. Altering these factors might boost the immune system and affect other areas of cancer biology, thereby allowing the chemotherapy to be more effective. The significance of this research is that it may help improve our treatments of this disease in the future.

ELIGIBILITY:
Preoperative Eligibility Criteria:

Inclusion Criteria

* Suspected preoperative diagnosis of invasive ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer based on imaging and CA-125 levels
* Patients must scheduled for a planned tumor debulking at least 72 hours in advance in order for the patient to take at least 48 hours of prescribed Propranolol
* Intention for chemotherapy administration at Washington University
* An approved informed consent and authorization permitting release of personal health information must be signed by patient or guardian
* Age ≥ 18 years
* Gynecologic Oncology Group performance status 0-2
* Patient's of childbearing age must have a negative pregnancy test

Exclusion Criteria

* Patients who receive neoadjuvant chemotherapy for their ovarian, primary peritoneal, or fallopian tube cancer are excluded.
* Patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated new invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer are eligible, provided that they have not received chemotherapy for any tumor
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation therapy for localized cancer of the breast, head and neck, or skin is permitted provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than stage IA; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesions.
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present with the last five years or whose previous cancer treatment contraindicates this protocol therapy are excluded.
* Use of systemic glucocorticoids such as Prednisone or Decadron in the last month
* Inability to accurately answer questions (e.g. dementia, brain metastases) or speak English
* Cirrhosis of the liver
* Patients with a GOG Performance status 3 or 4
* Patients under the age of 18
* Comorbid conditions: Addison's disease, autoimmune hepatitis, hepatitis B, hepatitis C, AIDS or HIV, lupus erythematosus, mixed connective tissue disease, rheumatoid arthritis
* Any patients already on beta-blockers or contraindicated to receive beta-blockers

Post-operative Eligibility Criteria:

Inclusion Criteria

* Histologic diagnosis of invasive epithelial ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer. Histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell carcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified. However, the histologic features must be compatible with primary Müllerian epithelial adenocarcinoma. Patients with low grade invasive epithelial ovarian cancers may participate.
* Stages I-IV of the above cancer
* Patients having undergone a suboptimal or optimal tumor debulking
* Gynecologic Oncology Group performance status 0-2
* Patients must have adequate:

  1. Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1500/ml.
  2. Platelets greater than 100,000/ml
  3. Renal function: Creatinine ≤ 1.5 x institutional upper limit normal
  4. Hepatic function: Bilirubin less than or equal to 1.5 x institutional upper limit normal; SGOT and alkaline phosphatase less than or equal to 2.5 x institutional upper limit normal.
  5. Neurologic function: Neuropathy (sensory and motor) less than or equal to grade 1 according to Common Toxicity Criteria for Adverse Events version 3 (CTCAE).
  6. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for the management of venous thrombosis including pulmonary embolus) and a PTT <1.2 times institutional upper limit of normal.

Exclusion Criteria

* Patients who have received targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their primary peritoneal, ovarian, or fallopian tube cancer. Patients cannot receive concurrent bevacizumab or other targeted therapy as part of their primary chemotherapy.
* Patients with non-epithelial ovarian tumors that do not require adjuvant chemotherapy, borderline epithelial ovarian tumor, or recurrent invasive epithelial ovarian, low grade ovarian cancer, primary peritoneal, or fallopian tube cancer treated with surgery only (such as patients with stage IA or IB)
* Patients with a synchronous primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than stage IA; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesions
* Metastases to the ovaries from other organs except fallopian tube or primary peritoneal carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of concurrent beta-blocker administration with chemotherapy | Completion of 6 cycles of chemotherapy/propranolol
  Proportion of patients who successfully complete 6 cycles of chemotherapy and concurrent treatment with propranolol

SECONDARY OUTCOMES:
Progression free survival rates | From time of diagnosis to 1 year following the 6th cycle of chemotherapy or 18 months following surgery
Pilot data on blood markers in patients with ovarian cancer pre- and post-beta blockade | Pre-surgery, Completion of 3rd cycle of chemo, Completion of 6th cycle of chemo
Characterization of biobehavioral states with surveys | Pre-surgery, Completion of 3rd cycle of chemo, Completion of 2nd cycle of chemo
  To characterize the biobehavioral states of these patients by using the Functional Assessment of Chronic Illness and Therapy- Ovary (FACT-O), Hospital Anxiety and Depression Survey (HADS) and the Center for Epidemiologic Studies Depression Scale (CESD)
Evaluation of immunohistochemistry of angiogenic markers on tumor samples | At time of initial surgery
  Immunohistochemistry for VEGF, IL-6, IL-8, MMP-2 and MMP-9 will be performed on tumor samples.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Thaker, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu